CLINICAL TRIAL: NCT06699329
Title: A Clinical Study to Evaluate the Effect of MK-0616 and Semaglutide on Their Respective Pharmacokinetics in Healthy Adult Participants
Brief Title: A Study of Enlicitide Decanoate (MK-0616) and Semaglutide in Healthy Adult Participants (MK-0616-023)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-023; MK-0616-023 (Other: MSD)
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enlicitide Decanoate and Semaglutide (Experimental): Period 1: Participants receive an oral dose of enlicitide decanoate every day for 1 week.
  Period 2: Participants receive an oral dose of semaglutide every day for 6 weeks.
  Period 3: Participants receive an oral dose of both enlicitide decanoate and semaglutide every day for 1 week.
  Interventions: Drug: Enlicitide Decanoate; Drug: Semaglutide

INTERVENTIONS:
Drug: Enlicitide Decanoate — multiple doses, oral tablet
  Other Names: MK-0616
Drug: Semaglutide — multiple doses, oral tablet
  Other Names: Rybelsus

SUMMARY:
The goal of this study is to learn what happens in a person's body over time when they take enlicitide decanoate and semaglutide alone or at the same time. Enlicitide decanoate is a new medicine that lowers the amount of cholesterol in a person's blood. Semaglutide is a drug used to treat type 2 diabetes.

Researchers want to learn what happens to the amount of semaglutide and enlicitide decanoate in a person's blood when each drug is taken alone and when they are taken together.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2
* Medically healthy with no clinically significant medical history

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* History of gastrointestinal disease which may affect food and drug absorption, or has had a gastric bypass or similar surgery
* History of cancer

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of Enlicitide Decanoate | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24hrs of enlicitide decanoate.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of Semaglutide | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24hrs of semaglutide.
Maximum Plasma Concentration (Cmax) of Enlicitide Decanoate | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Cmax of enlicitide decanoate.
Maximum Plasma Concentration (Cmax) of Semaglutide | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Cmax of semaglutide.
Time to Maximum Plasma Concentration (Tmax) of Enlicitide Decanoate | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Tmax of enlicitide decanoate.
Time to Maximum Plasma Concentration (Tmax) of Semaglutide | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Tmax of semaglutide.

SECONDARY OUTCOMES:
Number of Participants Who Experience a Treatment-Emergent Adverse Event (TEAE) | Up to approximately 12 weeks
  An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. The number of participants who experience a TEAE will be reported.
Number of Participants Who Discontinue Study Due to a TEAE | Up to approximately 12 weeks
  An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. The number of participants who discontinue study due to a TEAE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com